CLINICAL TRIAL: NCT04175366
Title: Shared Decision Making in Psychiatric Inpatient Care to Enhance Patient Participation
Brief Title: Shared Decision Making in Psychiatric Inpatient Care
Acronym: DEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DEAL2019UmU
Record Dates: First submitted 2019-11-14; First posted 2019-11-25 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-11

CONDITIONS: Participation, Patient; Psychiatric Hospitalization; Psychosis
Keywords: Shared Decision Making; Compulsory Care; Psychiatric Care
MeSH Terms: conditions — Patient Participation; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making (Experimental): Intervention with Shared Decision Making procedure regarding decision on planning of care and treatment before discharge.
  Interventions: Other: Shared Decision Making
- Care as usual (No Intervention): Discharge planning as usual.

INTERVENTIONS:
Other: Shared Decision Making — Shared Decision Making including adapted decision aid.
  Arms: Shared Decision Making

SUMMARY:
Introduction

National guidelines and The Patient Act from 2014 call for an active role for the patient in the decision making process. The role of the doctor is not only to give advice and to prescribe treatments, but also to present different alternatives with pros and cons. The method of Shared Decision Making (SDM) is meant to improve patient participation in line with ethical guidelines and legal demands. In summary, SDM consists of three steps:

1. To introduce a choice.
2. To discuss the options.
3. To make a shared decision. Systematic studies on SDM show patients becoming better informed and less uncertain regarding decisions made, and decisions closer to clinical guidelines compared to treatment as usual (TAU). It is still unresolved if SDM leads to improved clinical outcomes.

Aim

The aim of the study is to investigate outcomes of SDM carried out in psychiatric inpatient care: the patients' perceived participation (primary outcome) and health related outcomes (secondary).

Method

The decision situation in focus for this project is the planning of hospital discharge and future outpatient care. The participants are randomized to either SDM or TAU. Patient participation will be measured by questionnaires, interviews with patients and recorded decision talks. Clinical outcomes will be measured 12 months after discharge.

Preliminary results

A pilot study conducted in 2017-2018 clarified the feasibility of instruments and the intervention, and gave data for power estimation.

DETAILED DESCRIPTION:
TITLE

DEAL Shared Decision Making in psychiatric inpatient care to enhance participation and autonomy.

PURPOSE AND AIMS

The purpose is to investigate patients' participation and autonomy in psychiatric inpatient care and the potential of Shared Decision Making (SDM) to strengthen patients' participation in clinical decision making.

PRIMARY OUTCOME:

Does SDM improve patient participation?

SECONDARY OUTCOMES:

Does the use of SDM improve clinical outcomes (length of inpatient days, length of involuntary care, number of inpatient episodes and completed outpatient visits)?

Does outcomes of SDM relate to gender, socio-economical background, severity of disease, level of function, diagnosis and compulsory/voluntary care?

How does patients and doctors experience SDM in psychiatric inpatient care regarding discharge planning?

What are the ethical and legal implications of practicing SDM in Swedish psychiatric care?

SDM DEFINED

SDM as it will be pursued in this project consists of three steps: To introduce choice. To discuss the options. To make a shared decision.

SDM aims to help patients to explore personal preferences, make informed decisions and achieve active participation in the decision-making process. From the perspective of patient autonomy, SDM goes beyond mere informed consent. The practice of SDM is meant to empower the patient to active participation.

METHOD

SDM in psychiatric inpatient care will be evaluated in a randomized controlled trial with SDM vs treatment as usual (TAU). The decision studied is the planning of care in the process of discharge from hospital.

Quantitative methodology is used to measure the level of perceived participation and clinical outcomes. The qualitative parts of the study will focus on the process of implementing SDM in inpatient psychiatric care, and to identify ethically and legally complex situations in the use of SDM.

RECRUITMENT PROCESS

Informed consent will be obtained from all participants. The participants will be randomized to either SDM or TAU. The randomization is conducted by slots of 40 persons per ward (20 SDM and 20 TAU) by SPSS random number series.

RESEARCH QUESTIONS

The primary outcome of patient perceived participation (including the decision making process) will be answered quantitatively with the questionnaires Dyadic OPTION, SURE, Collaborate and SDM-Q-9, and qualitatively with interviews by phone 3 weeks after discharge. The interviews will be audio recorded and analyzed using qualitative content analysis. Perceived participation will be measured at inclusion at the ward and after the discharge planning conversation in both the SDM and TAU group with the questionnaires.

Clinical effects (secondary outcomes) will be studied by number of: inpatient days, days of compulsory care, inpatient episodes, completed outpatient visits, completed decisions and emergency visits one year after the discharge. Information will be obtained from clinical records.

Clinical and social factors will be related to level of participation. Data collected: gender, level of education, severity of illness (CGI-S), level of function (GAF) and voluntary/compulsory admission at inclusion, quality of life at discharge (EQ-5D) and clinical diagnosis at discharge (clinical records).

The patient-doctor decision talks will be recorded and analyzed using qualitative content analysis, focusing on ethical and legal questions.

STUDY PLAN

The study starts in the fall of 2019 with a short education for the doctors and staff at the wards in the form of a seminar on SDM in a recovery perspective. The written decision support, a step-by-step manual to facilitate SDM is used in role plays and simulations to prepare the staff. Patients receive an illustrated and easy-to-read information and decision guide.

During 2019-2021 patients will be recruited. This will include informed consent to participate in the study, to collect clinical data from medical records (12 months in retrospect and 12 months prospective from day of discharge), to recorded decision talks and to conduct a telephone interview three weeks after discharge.

Follow up data will be collected in 2021-2022, publication of results is planned in 2022.

DATA ANALYSIS

A power estimation based on the results of the pilot study with a power of 80% and an α error probability of 0.05 gave a Cohens d of 0,672.

G*Power was also used for an a priori estimation with a power of 80% and an α error probability of 0.05. A Cohen´s d of 0.5 was chosen since there is a greater risk of contamination between groups in the randomized study. This gave a group size of n=53 persons needed in each group. The dropout rate in the pilot study of 50% is with adjustments and new approaches still reasonable to estimate to approximately 30%. Group sizes were estimated to n=80 persons and the total inclusion number of N=160 persons.

The groups (SDM vs TAU) will be compared for difference in mean rank, using a Wilcoxon-Mann-Whitney test, regarding their perceived participation in the decision process, which is the primary outcome. For the secondary outcomes comparison between the two groups with t-tests, comparing means will include number of inpatient days, number of inpatient episodes, number of involuntary inpatients days and completed outpatient visits.

For other secondary outcomes, such as the relation between patient perceived participation and social/clinical factors, a multifactor analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* Admission to psychiatric inpatient care.
* Informed consent to study participation.

Exclusion Criteria:

* Lack of basic language skills in Swedish.
* Earlier enrollment in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient record.
Enrollment: 160 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Level of patient perceived participation | Measurement 6 weeks after inclusion or at discharge if earlier.
  Measurement with the questionnaire Dyadic OPTION, with a sum score of 1-44 where 44 is the highest perceived participation.
Level of patient perceived participation | Measurement 6 weeks after inclusion or at discharge if earlier.
  Measurement with the questionnaire SDM-Q-9 with a sum score of 0-45 where 45 is the highest perceived participation.
Level of patient perceived participation | Measurement 6 weeks after inclusion or at discharge if earlier.
  Measurement with the questionnaire Collaborate with a sum score of 0-12 where 12 is the highest perceived participation.
Level of patient perceived participation | Measurement 6 weeks after inclusion or at discharge if earlier.
  Measurement with the questionnaire SURE, (Sure of myself; Understand information; Risk-benefit ratio; Encouragement) screening test for decisional conflict in patients, with a sum score of 0-4 where 4 is the highest perceived participation.

SECONDARY OUTCOMES:
Percentage of carried out planned outpatient visits | 1 year
Number of rehospitalisations | 1 year
Days of compulsory care | 1 year
Number of episodes of compulsory care | 1 year
Number of inpatient days | 1 year
Number of emergency visits | 1 year
Days until rehospitalisation | 1 year
Percentage of decisions on social support carried out | 1 year
Level of quality of Life: EuroQol EQ-5D | Measurement 6 weeks after inclusion or at discharge if earlier.
  Measurement with the questionnaire EuroQol EQ-5D with a score of 0-1 where 1 is the highest quality of life.
Level of quality of Life: EuroQol EQ-VAS | Measurement 6 weeks after inclusion or at discharge if earlier.
  Measurement with the questionnaire EuroQol EQ-VAS with a score of 0-100 where 100 is the highest quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Sandlund, Professor, Principal Investigator — Umeå University
Locations (2):
- Sweden (2):
  - Ward 5, Stockholms Norra Psykiatri, Stockholm, Sverige
  - Ward 1 and 2, Umeå Psykiatri, Umeå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joosten EA, DeFuentes-Merillas L, de Weert GH, Sensky T, van der Staak CP, de Jong CA. Systematic review of the effects of shared decision-making on patient satisfaction, treatment adherence and health status. Psychother Psychosom. 2008;77(4):219-26. doi: 10.1159/000126073. Epub 2008 Apr 16. PMID 18418028
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Hamann J, Cohen R, Leucht S, Busch R, Kissling W. Shared decision making and long-term outcome in schizophrenia treatment. J Clin Psychiatry. 2007 Jul;68(7):992-7. doi: 10.4088/jcp.v68n0703. PMID 17685733
- [Background] Stovell D, Morrison AP, Panayiotou M, Hutton P. Shared treatment decision-making and empowerment-related outcomes in psychosis: systematic review and meta-analysis. Br J Psychiatry. 2016 Jul;209(1):23-8. doi: 10.1192/bjp.bp.114.158931. Epub 2016 May 19. PMID 27198483
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Slade M. Implementing shared decision making in routine mental health care. World Psychiatry. 2017 Jun;16(2):146-153. doi: 10.1002/wps.20412. PMID 28498575